CLINICAL TRIAL: NCT00108524
Title: A Low-Carbohydrate, Ketogenic Diet Versus Orlistat for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-005-03F
Record Dates: First submitted 2005-04-15; First posted 2005-04-18 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: anti-obesity agents; diet therapy; diet, reducing; obesity; overweight; risk factors; weight loss
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Overweight; Weight Loss | interventions — Orlistat; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Carbohydrate Ketogenic Diet (Experimental): Participants receive dietary counseling over 48 weeks aimed at helping them to lower starch and sugar intake.
  Interventions: Behavioral: Low carbohydrate ketogenic diet
- Low-Fat Diet plus Orlistat (Active Comparator): Participants receive counseling on a low fat diet over 48 weeks aimed at reducing fat and calorie intake, and additionally receive Orlistat taken 3 times daily.
  Interventions: Drug: Orlistat; Behavioral: Low-fat diet

INTERVENTIONS:
Behavioral: Low carbohydrate ketogenic diet — A low-carb diet limits carbohydrates - such as grains, starchy vegetables and fruit - and emphasizes dietary protein and fat.
  Arms: Low Carbohydrate Ketogenic Diet
Drug: Orlistat — In addition to the low fat diet, Orlistat is taken 3 times daily.
  Other Names: Xenical
  Arms: Low-Fat Diet plus Orlistat
Behavioral: Low-fat diet — Participants receive counseling on a low fat diet over 48 weeks aimed at reducing fat and calorie intake
  Arms: Low-Fat Diet plus Orlistat

SUMMARY:
This study compares two types of diet interventions: a low carbohydrate ketogenic diet (Atkins) and a low-fat diet combined with a medication (Orlistat).

DETAILED DESCRIPTION:
Overweight and obesity are increasingly prevalent in the veteran population as well as the general public. For patients with obesity-associated illnesses, there are few effective treatment options available after failed attempts at diet and exercise, even though weight loss has been shown to alleviate these conditions. The purpose of this study is to compare the tolerability, safety, and efficacy of a low-carbohydrate ketogenic diet (Atkins) with a combination of a low-fat diet and Orlistat. The outcomes examined over a 48 week duration will include body weight, risk factors for heart disease (e.g., lipid profiles), and blood sugar. This is a randomized, parallel-intervention trial. Subjects (n=150) will be recruited from the Durham VAMC Ambulatory Care Clinics. All patients receive one of the two intensive weight loss interventions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a VA medical center primary care provider;
* Failed first line diet and exercise recommendations;
* In stable health by screening physical and lab tests;
* Agrees to make regular visits per study protocol;
* Has access to telephone;
* Body mass index (BMI) > or = 27 with obesity-related illness OR BMI > or = 30 with no risk factors;
* No contraindications to Orlistat;
* Not pregnant or breast-feeding;
* No serious mental health illness such as dementia or schizophrenia;
* No use of a weight loss therapy in the month prior to screening.

Exclusion Criteria:

* No VAMC primary care provider
* Unable to attend regular study visits
* No access to telephone
* BMI < 27
* Contraindications to Orlistat
* Pregnancy, breast feeding or planning to become pregnant
* Unstable mental health illness
* Use of a weight loss therapy in the month prior to screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2004-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William S. Yancy, MD MHS, Principal Investigator — Durham VA Medical Center HSR&D COE
Locations (1):
- Durham VA Medical Center HSR&D COE, Durham, North Carolina, United States

REFERENCES:
- [Result] Mayer SB, Jeffreys AS, Olsen MK, McDuffie JR, Feinglos MN, Yancy WS Jr. Two diets with different haemoglobin A1c and antiglycaemic medication effects despite similar weight loss in type 2 diabetes. Diabetes Obes Metab. 2014 Jan;16(1):90-3. doi: 10.1111/dom.12191. Epub 2013 Aug 29. PMID 23911112
- [Result] Yancy WS Jr, Almirall D, Maciejewski ML, Kolotkin RL, McDuffie JR, Westman EC. Effects of two weight-loss diets on health-related quality of life. Qual Life Res. 2009 Apr;18(3):281-9. doi: 10.1007/s11136-009-9444-8. Epub 2009 Feb 11. PMID 19212822
- [Result] Yancy WS Jr, Westman EC, McDuffie JR, Grambow SC, Jeffreys AS, Bolton J, Chalecki A, Oddone EZ. A randomized trial of a low-carbohydrate diet vs orlistat plus a low-fat diet for weight loss. Arch Intern Med. 2010 Jan 25;170(2):136-45. doi: 10.1001/archinternmed.2009.492. PMID 20101008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient clinics affiliated with the Department of Veterans Affairs Medical Center in Durham, North Carolina, between April 2005 and October 2006.
Pre-assignment Details: 18-70yo,BMI 27-30+obesity-related disease or BMI>30 regardless of comorbidity. Excluded:weight loss in <30 days;pregnant,breastfeeding,DM-1;unstable heart disease or psych illness,dementia,substance abuse;HTN >160/100; creatinine>1.5men,>1.3women; HemA1c>11%; triglyceride>600; LDL-C>190. Not considered enrolled if not told group assignment (n=14).
Groups:
- Low Carbohydrate Ketogenic Diet: Participants receive dietary counseling over 48 weeks aimed at helping them to lower starch and sugar intake.
  Low carbohydrate ketogenic diet: Participants were instructed to restrict carbohydrate intake initially to less than 20 g/d using pocket guides and handouts. Participants could eat unlimited meat and eggs, 112 g of hard cheese, 0.48 L of low-carbohydrate vegetables (eg, leafy greens), and 0.24 L of moderate-carbohydrate vegetables (eg, broccoli, asparagus) daily; calorie intake was not restricted. As participants approached their goal weight or if cravings threatened their adherence to the diet, they were advised to add approximately 5 g of carbohydrates to their daily intake each week until weight was maintained or cravings diminished.
- Low-Fat Diet Plus Orlistat: Participants receive dietary counseling over 48 weeks aimed at reducing fat and calorie intake and additionally receive Orlistat taken 3 times daily.
  Orlistat plus a low-fat diet: Participants were instructed to restrict intake of total fat (<30% of daily energy), saturated fat (<10% of daily energy), cholesterol (<300 mg daily), and calories using pocket guides, handouts, and individualized goals. Recommended calorie intake was 500 to 1000 kcal below a participant's calculated weight maintenance intake. In addition, a 30-day supply of orlistat (120 mg before meals 3 times a day) was provided monthly.
Period: Overall Study
Arm/Group | Low Carbohydrate Ketogenic Diet | Low-Fat Diet Plus Orlistat
Started | 81 | 79
Completed | 52 | 61
Not Completed | 29 | 18

BASELINE CHARACTERISTICS:
Population: 160 participants were randomized (81 allocated to LCKD, 79 to Orlistat plus LFD). 14 did not receive the intervention. 33 discontinued the intervention. Out of the 146 participants analyzed, 113 completed the intervention.
Groups:
- Arm 1: Participants receive dietary counseling over 48 weeks aimed at helping them to lower starch and sugar intake.
  Low carbohydrate ketogenic diet: Participants were instructed to restrict carbohydrate intake initially to less than 20 g/d using pocket guides and handouts. Participants could eat unlimited meat and eggs, 112 g of hard cheese, 0.48 L of low-carbohydrate vegetables (eg, leafy greens), and 0.24 L of moderate-carbohydrate vegetables (eg, broccoli, asparagus) daily; calorie intake was not restricted. As participants approached their goal weight or if cravings threatened their adherence to the diet, they were advised to add approximately 5 g of carbohydrates to their daily intake each week until weight was maintained or cravings diminished.
- Arm 2: Participants receive dietary counseling over 48 weeks aimed at reducing fat and calorie intake and additionally receive Orlistat taken 3 times daily.
  Orlistat plus a low-fat diet: Participants were instructed to restrict intake of total fat (<30% of daily energy), saturated fat (<10% of daily energy), cholesterol (<300 mg daily), and calories using pocket guides, handouts, and individualized goals. Recommended calorie intake was 500 to 1000 kcal below a participant's calculated weight maintenance intake. In addition, a 30-day supply of orlistat (120 mg before meals 3 times a day) was provided monthly.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 72 | 74 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 74 | 146
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (10.2) | 52.0 (9.2) | 52 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 52 | 53 | 105
Region of Enrollment [Number; unit: participants]
  United States | 72 | 74 | 146

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight at 48 Weeks
Description: Body weight was measured using the same calibrated scale (Tanita Corp, Arlington Heights, Illinois) at each visit at the same time of day, with the participant wearing light clothing and no shoes.
Time Frame: baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: percentage of weight loss
Groups:
- Arm 1: Low carbohydrate ketogenic diet: Participants receive dietary counseling over 48 weeks aimed at helping them to lower starch and sugar intake.
- Arm 2: Orlistat plus a low-fat diet: Participants receive dietary counseling over 48 weeks aimed at reducing fat and calorie intake and additionally receive Orlistat taken 3 times daily.
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 72 | 74
percentage of weight loss | -9.5 [-14.8 to -7.9] | -8.5 [-11.0 to -6.1]

2. Secondary Outcome: Change From Baseline in Risk Factors for Heart Disease (e.g., Lipid Profiles) at 48 Weeks
Description: Measured change in low-density lipoprotein cholesterol, or LDL-C, from baseline to 48 weeks.
Time Frame: baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 72 | 74
mg/dL | -1.91 [-8.14 to 4.33] | -8.29 [-14.06 to -2.52]

3. Secondary Outcome: Change From Baseline in Blood Sugar at 48 Weeks
Description: Measured change in Fasting glucose, mg/dL, from baseline to 48 weeks.
Time Frame: Baseline and 48 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 72 | 74
mg/dL | -9.74 [-16.93 to -2.55] | -3.54 [-10.05 to -3.26]

ADVERSE EVENTS:
Time Frame: 48 weeks
Description: The O + LFD participants reported gastrointestinal effects more frequently than the LCKD participants, occurring predominantly after dietary indiscretions. The LCKD had its own gastrointestinal adverse effect, constipation, in most cases resolving by increasing fluid and dietary fiber intake and/or adding a fiber supplement or stool softener.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 1/72 | 2/74
Other Adverse Events (participants affected / at risk) | 49/72 | 30/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=72) | Arm 2 (N=74)
gastrointestinal symptoms (Gastrointestinal disorders) | 1 (1) | 2 (2) — 1 participant discontinued orlistat treatment due to intolerance of gastrointestinal symptoms.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=72) | Arm 2 (N=74)
constipation (Gastrointestinal disorders) | 49 (49) | 30 (30) — constipation

LIMITATIONS AND CAVEATS:
We provided orlistat at no cost. This could have increased dietary adherence, attendance, and/or retention compared with the LCKD and may lead to different results than what might be seen in patients who must pay for orlistat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes